CLINICAL TRIAL: NCT06680856
Title: Phase II, Multicenter, Double Blind, Randomized Controlled Trial on "Off the Shelf" Allogeneic Platelet Rich Plasma (PRP) to Treat Diabetic Foot Ulcers
Brief Title: Allogeneic Platelet Rich Plasma (PRP) to Treat Diabetic Foot Ulcers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ospedale Policlinico San Martino (Other)
Collaborators: IRCSS Istituto Dermopatico dell'Immacolata, Fondazione Luigi Maria Monti (Other); Universita degli Studi di Genova (Other)
Responsible Party: Principal Investigator, Giovanni Pratesi, MD, Professor in Vascular Surgery, Ospedale Policlinico San Martino
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RF-2018-12366868
Record Dates: First submitted 2024-10-31; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Foot Ulcer; Skin Lesions; Allogeneic; PRP
Keywords: allogeneic Platelet Rich Plasma; diabetic foot ulcer; Hyaluronic acid; skin regeneration
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: * Experimental Group: Platelet Rich Plasma + Hyaluronic Acid (PRP+HA) (Group 1)
  * Control Group: Hyaluronic acid gel (HA) (Group 2)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP+HA (Experimental): Diabetic foot ulcers were treated with PRP+HA dressing
  Interventions: Combination Product: PRP+HA
- HA alone (Active Comparator): Diabetic foot ulcers were treated with HA dressing alone
  Interventions: Combination Product: HA

INTERVENTIONS:
Combination Product: PRP+HA — treatment of diabetic foot ulcers with allogeneic PRP+HA
  Arms: PRP+HA
Combination Product: HA — treatment of diabetic foot ulcers with HA
  Arms: HA alone

SUMMARY:
Chronic skin ulcers pose a major health burden because of population aging and increased prevalence of chronic diseases such as diabetes. Standard therapy, such as ulcer debriding and physical treatments, is in most cases palliative. Autologous Platelet Rich Plasma (PRP) as enhancer of healing was proposed as a real innovation in the field. However, conflicting results were obtained by different groups, because of the different production and clinical protocols and inter-individual variability in the patient's blood.

A multi center double-blind, randomized clinical trial was conducted to test an allogeneic platelet-derived product obtained from large pools of blood donations for the treatment of diabetic foot ulcers in association with Hyaluronic Acid (HA) dressing as compared to Hyaluronic Acid alone. Being prepared in batches, the product undergoes rigorous Quality Control analysis before use. An allogeneic PRP product would represent a substantial improvement in the treatment of skin ulcers.

DETAILED DESCRIPTION:
Background Skin ulcers are open sores often accompanied by the sloughing-off of inflamed tissue. Chronic skin ulcers pose a major global health burden since they are closely linked to population aging and chronic diseases such as diabetes . There is a strong association between pain and quality of life, which are worse for larger ulcers with longer duration. Women have both more pain and poorer quality of life than men. Chronic skin ulcers recur frequently and heal poorly. 1/5 ulcers are still not healed after 2 years, and 1/12 are still open after 5 years and can last more than 10 years. Diabetes is the most common cause of ulcers in Europe and the USA. Diabetic patients have a lifetime risk of foot ulcer as high as 25%. Non healing chronic ulcers of the lower limbs in patients with type 1 or 2 diabetes are at increased risk of complications, including infections and amputation. Approximately 50% of diabetic foot ulcers become infected, and 20% of these require amputation .

Chronic skin ulcers are difficult to treat also because of impaired blood flow and infection. Present standard treatment of diabetic ulcers includes regular debridement, off-loading, treatment of infection, revascularization when appropriate,optimizing metabolic control, and the treatment of any concomitant diseases, as well as education about foot care and the provision of appropriate footwear. However, healing rates are highly variable, and recurrences frequent .

Autologous Platelet Rich Plasma (PRP) to treat chronic skin ulcers through the reactivation of dormant endogenous regeneration mechanisms is truly innovative. In fact, PRP not only increases endothelial cells recruitment and improves vascularization, but also promotes recruitment of macrophages which, in turn, through their paracrine activity, recruit and stimulate proliferation of mesenchymal and epithelial stem/progenitor cells, leading to synthesis of extracellular matrix molecules and skin regeneration. There is clinical evidence that autologous PRP gel therapy improves healing of chronic skin ulcers, but treatment of diabetic ulcers by autologous PRP is often hampered because diabetes leads to a reduced and/or inadequate production of growth factors, angiogenic response, impaired function of macrophages, reduced formation of granulation tissue, abnormal migration, and proliferation of fibroblasts and keratinocytes.

Moreover, before this new therapeutic approach can be available to a large population of patients, several issues need to be addressed. While some groups reported encouraging results on PRP as enhancer of tissue healing, others failed to observe an improvement in the healing process. This may be due to a poor quality of the PRP. In fact, there is significant inter-individual variability in platelet concentration, which can significantly vary depending on the health status of the different patients. Variability also exists in preparations from different Centers. In many cases, PRP is prepared based on non-standardized protocols, or by using commercially available devices that may be not fully adequate. Further limitations include difficulty to obtain sufficient quantities of blood from the elderly, or from debilitated patients with limited mobility, as well as the lack of prompt PRP availability, and the high production cost.

Hyphothesis and Significance:

The use of allogeneic PRP, obtained from a pool of blood donations, would be advantageous over the use of autologous PRP, and could be the only alternative when the autologous PRP is not available.

This multicenter clinical trial tested an allogeneic platelet-derived product, obtained from pools of blood donations according to standardized large-scale procedures. This product would represent a substantial improvement in the treatment of chronic skin ulcers. Furthermore, allogeneic PRP - produced in batches and not immediately used underwent a rigorous Quality Control analysis before its clinical use.

Specific Aim 1:

Implementation of a phase II, multicenter, double-blind, randomized controlled trial on "off the shelf" allogeneic PRP to treat diabetic foot ulcers. The protocol was approved by the pertinent Ethical Committees prior to project start.

The trial was conducted in accordance with the protocol and in compliance with European and local legal and regulatory requirements, as well as the general principles set forth in the Guidelines for Good Clinical Practice (CPMP/ICH/135/1995) and the Declaration of Helsinki (World Medical Association - 2013).

The primary aim of this study was to evaluate whether allogeneic PRP could improve the rate of healing of foot ulcers in diabetic patients. Preparations of allogeneic PRP in association with hyaluronic acid dressing were compared with hyaluronic acid only.

The primary endpoint is the cumulative rate of wound healing at the end of the 12 week follow-up.

Patients were randomized in a 1:1 ratio to:

* Experimental Group: Treatment with offloading, debridement, and hyaluronic acid gel + PRP gel;
* Control Group: Treatment with offloading, debridement, and hyaluronic acid gel

Specific Aim 2:

Secondary aim was the evaluation of the safety of the allogeneic PRP.

Specific Aim 3:

Third aim was to study the immune response after allogeneic PRP treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females
2. Between the ages of 40 and 90 years
3. Diagnosis of diabetes: random glycaemia >126 mg in more sample or second hour oral Glucose Tolerance Test glycaemia >200 mg or glycosylated hemoglobin >6.5 mmol/L
4. The cross-sectional area of the index ulcer will be between 25 and 2000 mm2
5. Injury-trophic level Grade I, II, Level A and B (according to Texas classification)
6. Ankle Brachial Index >0.5
7. The patient's willingness to cooperate with the physician in follow-up
8. No previous treatment with platelet derivatives
9. Negative serum pregnancy test within 7 days prior to commencement the treatment in premenopausal women.
10. Fertile women must use an effective method of contraception during the treatment and for at least 6 months after completion of treatment as directed by their physician.
11. Signature of the informed consent form

Exclusion Criteria:

1. Have End-Stage Renal Disease (ESRD-stage 5 of kidney disease), or severe heart failure which may require organ transplantation
2. Are breast-feeding.
3. Have a previous or current history of malignant neoplastic disease within the past 5 years
4. Have neuropsychiatric diseases that may interfere with the patient's ability to collaborate in the study.
5. They have any condition that, in the doctor's judgment, could endanger them.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
wound size measurements of diabetic foot ulcer lesion | 12 weeks
  The cumulative rate of wound healing at the end of the 12 week follow-up was determined by computed-aided imaging on standard pictures of the lesion taken at different times

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 0,1,2,3,4 and 12 weeks
  Incidence of Adverse Events at any site classified according to the Common Toxicity criteria of Adverse Events e.g. pain, disability, stress, etc.)

OTHER OUTCOMES:
measurement of HLA antigens in PRP treated patient | 0,4,12 weeks
  investigate formation of antibodies against donor HLA antigens by the recipient to study the immune response after allogeneic PRP treatment

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Pratesi, MD, Principal Investigator — IRCCS Ospedale San Martino
Locations (2):
- Italy (2):
  - IRCCS Ospedale San Martino, Genova, GE
  - Istituto dermatopatico dell'Immacolata, Roma

IPD SHARING:
Plan to Share IPD: No